CLINICAL TRIAL: NCT05273333
Title: Effect of Ultra-gyn® on Vulvovaginal Candidiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SbO216
Record Dates: First submitted 2022-02-09; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Vulvovaginal Candidiasis, Genital
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Intervention Model Description: A Prospective, Single-center, Open-label, Post-market Clinical Follow-up Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultra-gyn® (Other): ovule
  Interventions: Device: Ultra-gyn®

INTERVENTIONS:
Device: Ultra-gyn® — Ultra-gyn® ovule intravaginal application, every evening before bedtime for a 10 days period.

SUMMARY:
The aim of this post-market clinical follow up study is to confirm the performance and the safety of Ultra-gyn® (when used in accordance with its approved labelling)

ELIGIBILITY:
Inclusion Criteria:

To be eligible, each patient must satisfy the following criteria:

1. Is a non-menopausal woman aged 18 to 45 years,
2. Suffering from a vulvovaginal candidiasis (according to clinical examination),
3. Who was being prescribed standard antifungal therapy for Vulvovaginal Candidiasis,
4. Has regular menstrual cycles (21-35 days) or no menstruation due to continuous use of contraception,
5. Is able to understand the study related information and to give a written informed consent,
6. Has signed the informed consent form before beginning any study procedure,
7. Agrees not to use other vaginal products than those planned in the study protocol, during participation in the study,
8. Agrees not to use a diaphragm, spermicide or latex condoms, contraceptive creams and spermicide ovules during participation in the study,
9. Uses an effective method of contraception (contraceptive steroid [oral, patch, injection, implant], intrauterine device, vasectomized partner, history of permanent sterilization such as tubal ligation, hysterectomy, etc.) or abstinence,
10. Has no condition that may interfere with the study assessments
11. Is affiliated to a health social security system,
12. Is able to comply with protocol requirements and respect the conditions of the study,

Exclusion Criteria:

Patients meeting at least one of the following criteria cannot be included in the study:

Criteria related to a medical condition that would compromise patient safety or data fidelity:

1. Has had a sexually transmitted disease in the 21 days preceding screening or detected on this occasion,
2. Has a history of recurrent fungaemia,
3. Has a history of recurrent vulvovaginal candidiasis (defined as more than four episodes of vulvovaginal candidiasis in the previous year or two episodes in the last six months),
4. Has had pelvic surgery in the 3 months prior to screening,
5. Has had uterine or vaginal bleeding of unknown etiology,
6. Immunocompromised,
7. Has any other severe chronic or acute medical or psychiatric condition that in the judgment of the Investigator, could interfere with the study assessments,
8. Is pregnant (positive pregnancy test at screening), has given birth less than 2 months ago or is breastfeeding,
9. Has changed her method of contraception in the 2 months prior to screening,

   Criteria related to contraindications to the product used within the study:
10. With a known allergy or presenting an hypersensitivity to one of the component of the study product,
11. Presenting a contraindication or special warning to the study product, according to the package leaflet, including concomitant use of antifungal therapy during Ultra-gyn application,

    Criteria related to medications or situations that would interfere with or compromise data fidelity
12. Has taken systemic or intravaginal antibiotic or antifungal agents (other than those prescribed during the inclusion visit) in the 14 days preceding the screening visit,
13. Is not willing to stop taking probiotics dietary supplements and food products enriched with probiotics,
14. Is planning to change her usual habits (hygiene, dietary habits, tobacco and alcohol consumption, physical activity and sexual life) during the study,
15. Has participated in an interventional clinical study in the month prior to inclusion.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of Ultra-gyn® in relieving the symptoms of Vulvovaginal Candidiasis | Day 0 to Day 30 (+/-5)
  Change in vulvovaginal symptoms (5-point rating scale (ranging from 0 to 4, where 0=None and 4=Very severe) for vaginal itching, vaginal burning or soreness and vaginal discharge)

SECONDARY OUTCOMES:
To assess the effect of Ultra-gyn® on Candida spp | Day 0 and Day 30 (+/-5)
  Change in vaginal load of Candida spp (CFU Enumeration)
To assess the effect of Ultra-gyn® on vaginal microbiota | Day 0 and Day 30 (+/-5)
  Analysis with shotgun metagenomic sequencing of change in taxonomic composition of the vaginal microbiota
To assess the incidence of adverse effects | Day 1 to Day 30 (+/-5)
  Number, nature and characteristics of any adverse reactions
To assess the incidence of device deficiencies | Day 1 to Day 30 (+/-5)
  Number, nature and characteristics of any device deficiencies

CONTACTS AND LOCATIONS:
Locations (1):
- IR, Quatre Bornes, Mauritius

IPD SHARING:
Plan to Share IPD: No